CLINICAL TRIAL: NCT03742011
Title: Health of Offspring Born to Mothers With Polycystic Ovary Syndrome in Guangzhou Cohort Study
Brief Title: Offspring Born to Mothers With Polycystic Ovary Syndrome in Guangzhou Cohort Study
Acronym: PCOS-BIG
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Principal Investigator, Xiu Qiu, Director of the Born in Guangzhou Cohort Study, Guangzhou Women and Children's Medical Center
Other Study IDs: 2018101502
Record Dates: First submitted 2018-10-29; First posted 2018-11-15 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: PCOS; Offspring, Adult; Hyperandrogenism; Epigenetics; Insulin Resistance; Endocrine Disorder; Metabolic Disturbance
Keywords: PCOS; Hyperandrogenism; Epigenetics; Glucolipid metabolism disorder
MeSH Terms: conditions — Hyperandrogenism; Insulin Resistance; Endocrine System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During pregnancy: maternal blood, urine and stool. At delivery: cord, cord blood and placenta. During Infancy：dry blood spot, stool and blood. During childhood:blood, buccal swab and stool.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Offspring Born to Mothers with Polycystic Ovary Syndrome in Guangzhou Cohort study (PCOS-BIG) was established to investigate the short- and long-term effects of intrauterine exposure to maternal PCOS on the health of offspring in Guangzhou, China. Data are collected regarding maternal PCOS subtypes, nursing, diet and education as well as health outcomes in their later life. Biological samples including blood and tissue samples are also collected from participants.

DETAILED DESCRIPTION:
According to preliminary survey, the prevalence of polycystic ovary syndrome (PCOS) among Chinese women reached 7.5%. Hyperandrogenism and insulin resistance were considered as the main pathogenesis of PCOS. As reported, the secretion of androgen is higher among women with PCOS than the healthy reference population throughout their fertile lives. Worth of concern, offspring of PCOS patients presented with glucolipid metabolism disorders as early as during their childhood, while whose pathogenesis remains unclear. Prenatal exposure of rhesus monkey in pregnant to androgens produces glucolipid metabolic alterations in offspring resembling those in PCOS, suggesting that the exposure of the fetus to hyperandrogenism during gestation could affect the glucolipid metabolism of PCOS offspring. Growing evidence shows that different exposures during pregnancy will affect the DNA methylation of offspring and disturb their endocrine and metabolism. A birth cohort would provide an opportunity to examine the short- and long-term effects of PCOS exposure, such as hyperandrogenism, on health consequences of the offspring.

ELIGIBILITY:
Inclusion Criteria:

* Offspring born to women diagnosed with PCOS
* Offspring born to women with <20 weeks of gestation, intended to eventually deliver in Guangzhou Women and Children's Medical Center
* Permanent residents or families intended to remain in Guangzhou for ≥3 years

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Offspring born to women diagnosed with PCOS
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values (Glucolipid metabolism disorders) | An average of 3 years old
  Participants with one or more abnormal laboratory values will be considered as with glucolipid metabolism disorder.

SECONDARY OUTCOMES:
Prevalence of gestational diabetes, pregnancy induced hypertension, and cesarean section | From the recruitment (≤ 20 weeks of gestation) to delivery
  Assessed by self-reported time of onset and electronic medical records
Prevalence of stillbirth, preterm birth, small for gestational age, large for gestational age and birth defect | At delivery
  Assessed by electronic medical records
Epigenetic profiles of offspring | At birth
  Profiling DNA methylation and histone acetylation etc., using cord blood samples
Weight changes | At birth, age of 6 weeks, 6 months, 1 year, 3 years, 6 years, 12 years and 18 years old
  Weight changes from birth, to age of 6 weeks, 6 months, 1 year, 3 years, 6 years, 12 years and 18 years old
Height changes | At birth, age of 6 weeks, 6 months, 1 year, 3 years, 6 years, 12 years and 18 years old
  Height changes from birth, to age of 6 weeks, 6 months, 1 year, 3 years, 6 years, 12 years and 18 years old
Change of intestinal flora | At age of 6 weeks, 6 months, 1 year, 3 years, 6 years, 12 years and 18 years old
  Assessed by analyses of stool samples
Neurodevelopment at early childhood | At age of 1 year old
  Assessed using Gesell Developmental Schedules, including five items of adaptive, gross motor, fine motor, language, and social function
Changes of the percentage of body fat | At age of 3 years,6 years, 12 years and 18 years old
  Assessed using Dual Energy X-Ray Absorptiometry
Screen of intelligence quotient of offspring | At age of 6 years old
  Assessed using Peabody Picture Vocabulary Test (PPVT) and Raven's Standard Progressive Matrices (SPM). Of whom the score of PPVT ≥ 85 and the score of SPM ≥ 90, the child will be considered as normal level of intelligence quotient and of whom the score of PPVT under 85 or the score of SPM under 90 will be considered as suspected lower intelligence quotient.
Intelligence quotient of offspring assessed by WPPSI-IV | At age of 6 years old
  Child screened as of suspected lower intelligence quotient will be assessed by Wechsler Preschool and Primary Scale of Intelligence-Fourth edition (WPPSI-IV), including 5 items: verbal comprehension, visual spatial, fluid reasoning, working memory and process speed. Scores of the five items are added to get the total score.
Number of Participants With Abnormal Laboratory Values (Glucolipid metabolism disorders) | At age of 6 years, 12 years and 18 years old
  Participants with one or more abnormal laboratory values will be considered as with glucolipid metabolism disorder.
Number of participants with reproductive endocrine disorders | At age of 12 years and 18 years old
  Assessed by assay of hormones, including follicle stimulating hormone (FSH), luteinizing hormone (LH), estradiol (E2), total testosterone (TT), free testosterone (FT), androstenedione (A4), dehydroepiandrosterone sulfate (DHEA-S) and sex hormone binding globulin (SHBG), and by acne scoring and hirsutism scoring (modified Ferriman-Gallway scoring system). Participants with one or more abnormal laboratory values, and/or acne score ≥ 1, and/or hirsutism score ≥ 5 will be considered as with reproductive endocrine disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Qiu, PhD, Principal Investigator — Guangzhou Women and Children's Medical Center, China
Locations (1):
- Guangzhou Women and Children's Medical Center, China, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou Z, Li R, Qiao J. Androgen profile in Chinese women with polycystic ovary syndrome in their reproductive years. Reprod Biomed Online. 2017 Sep;35(3):331-339. doi: 10.1016/j.rbmo.2017.05.019. Epub 2017 Jun 16. PMID 28684272
- [Result] Qiu X, Lu JH, He JR, Lam KH, Shen SY, Guo Y, Kuang YS, Yuan MY, Qiu L, Chen NN, Lu MS, Li WD, Xing YF, Zhou FJ, Bartington S, Cheng KK, Xia HM. The Born in Guangzhou Cohort Study (BIGCS). Eur J Epidemiol. 2017 Apr;32(4):337-346. doi: 10.1007/s10654-017-0239-x. Epub 2017 Mar 20. PMID 28321694